CLINICAL TRIAL: NCT02222142
Title: Comparison of Propofol and Isoflurane Anesthesia on Cardioprotection and Clinical Outcomes in Patients Undergoing Off-pump Coronary Artery Bypass Graft Surgery : A Propensity-score Analysis
Brief Title: Volatile Versus Propofol Anesthesia in OPCAB
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Jong Hwan Lee, Assistant professor, Samsung Medical Center
Other Study IDs: 2013-09-127
Record Dates: First submitted 2014-08-17; First posted 2014-08-21 (Estimated); Last update posted 2014-08-21 (Estimated); Status verified 2014-08

CONDITIONS: Off Pump Coronary Artery Bypass Graft
Keywords: Ischemic heart disease; Off pump coronary artery bypass graft; Isoflurane; Propofol
MeSH Terms: conditions — Myocardial Ischemia | interventions — Isoflurane

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Isoflurane group: Isoflurane inhalational anesthesia during OPCAB
  Interventions: Drug: Isoflurane
- Propofol group: Total intravenous anesthesia with propofol during OPCAB

INTERVENTIONS:
Drug: Isoflurane — Comparison between isoflurane and propofol, Retrospective study
  Other Names: inhalational anesthetics
  Groups: Isoflurane group

SUMMARY:
Off pump coronary artery bypass graft (OPCAB) still requires myocardial protection owing to intermittent regional ischemic episode. The investigators retrospectively evaluated the cardioprotective and clinical outcomes of propofol versus isoflurane anesthesia in patients undergoing OPCAB.

DETAILED DESCRIPTION:
Several experimental and clinical researches have suggested that volatile anesthetics may reduce mortality in cardiac surgery owing to its preconditioning induced cardioprotective effect. Off-pump coronary artery bypass graft (OPCAB) surgery still requires cardioprotective strategies due to coronary hypoperfusion during anastomosis. The aim of this study was to evaluate the possible cardioprotective effect and clinical outcomes of propofol versus isoflurane anesthesia in patients undergoing OPCAB using propensity matching.

ELIGIBILITY:
Inclusion Criteria:

* OPCAB

Exclusion Criteria:

* On pump conversion

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients underwent OPCAB from January, 2010 to December, 2012
Sampling Method: Non-Probability Sample
Enrollment: 1080 (Actual)
Dates: Start 2010-01; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
CK-MB, CRP | Change from preoperative value in CK-MR and CRP at Postoperative day(POD), POD 1 and 2
  Comparison of CK-MB and CRP values between propofol and isoflurane groups on postoperative day, POD1 and POD 2

SECONDARY OUTCOMES:
Clinical adverse outcomes | until 1 year after OPCAB
  clinical adverse outcomes until postoperative 1 year

OTHER OUTCOMES:
Cardioprotection and clinical adverse outcomes in diabetic patients | POD, POD 1, POD 2, one month, one year
  primary and secondary outcome analysis in diabetic patients

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung medical center, Seoul, South Korea